CLINICAL TRIAL: NCT03522181
Title: Glucose-insulin-potassium Therapy Improves Lactic Acidosis in Liver Transplantation
Acronym: GIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central South University (Other)
Responsible Party: Principal Investigator, Ru-Ping Dai, professor, Central South University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XYEYYCT2016214
Record Dates: First submitted 2016-12-01; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Liver Transplantation
MeSH Terms: interventions — Sodium Chloride; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- control group (Placebo Comparator): saline
  Interventions: Other: saline
- GIK group (Experimental): glucose-Insulin-Potassium(GIK) infusion
  Interventions: Other: Insulin

INTERVENTIONS:
Other: saline — saline
  Arms: control group
Other: Insulin
  Other Names: glucose-Insulin-Potassium(GIK) infusion
  Arms: GIK group

SUMMARY:
Lactic acidosis is a common phenomenon occurring during orthotopic liver transplantation (OLT), especially during the anhepatic and early postreperfusion phases. However, little drugs effectively decrease the degree of lactic acidosis when it happens. The aim of this study is to explore whether glucose-Insulin-Potassium(GIK) infusion can relieve metabolic acidosis and improve perioperative outcome in patients undergoing OLT.

DETAILED DESCRIPTION:
Intraoperative metabolic acidosis begins soon after graft reperfusion and persists for several days. The current standard treatment for severe acidosis during OLT is NaHCO3, although it may compromise myocardial performance, exacerbate lactic acid accumulation and cause central nervous system demyelination. Surgical procedure is a primary source of endogenous lactic acid production, especially visceral ischemia originating from anhepatic stage. The present study thus hypothesized that GIK solution may improve metabolic acidosis in OLT patients through its unique effects of metabolic alleviation. Patients for orthotopic liver transplantation was enrolled and received either GIK or placebo. GIK or placebo infusion started after anesthesia induction. Intraoperative measures were mean arterial pressure, HR, arterial blood gases, lactate, glucose, Na, liver and renal function indexes. Outcome measures were time to tracheal extubation, intensive care unit, length of stay, complications, hospital length of stay, requirement for postoperative plasma transfusion, retransplantation, and perioperative mortality.

ELIGIBILITY:
Inclusion Criteria:

* patients who were to undergo OLT

Exclusion Criteria:

* diabetes mellitus, hyperkalemia on arrival (K+ > 5.5 mEq/L) and the inability to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02; Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
degree of lactic acidosis | up to 1 weeks
  Blood samples for arterial blood pH, PCO2 , PO2 , base excess, hematocrit, and plasma concentrations of lactic acid and Na were analyzed

OTHER OUTCOMES:
tracheal extubation | up to 3 days
  The time of tracheal extubation was calculated.
intensive care unit length of stay and hospital length of stay | up to 1 month
  The intensive care unit length of stay and hospital length of stay was calculated
The incidence of complications | up to 1 month
  The incidence of complications including liver dysfunction, renal dysfunction, infection, was analyzed
The incidence of retransplantation | up to 1 month
  The incidence of liver retransplantation
The incidence of perioperative mortality | up to 1 month
  The incidence of perioperative mortality

CONTACTS AND LOCATIONS:
Overall Officials: Ru-Ping Dai, MD, Principal Investigator — Second Xiangya Hospital of Central South University
Locations (1):
- Department of Anesthesiology, The Second Xiangya Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided